CLINICAL TRIAL: NCT02689687
Title: Automated Hovering to Improve Medication Adherence and Weight Management Among Congestive Heart Failure Patients: A Pilot Study
Brief Title: Automated Hovering for Congestive Heart Failure Patients: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 824067; 1R01HL128465-01 (NIH)
Record Dates: First submitted 2016-01-28; First posted 2016-02-24 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All participants will be (1) given an electronic pill bottle for their diuretic and a Bluetooth scale; (2) asked to provide the coordinator with name and contact information of a family member or friend to serve as a support partner; (3) will be assigned a 2-digit number to be used as part of the lottery-based engagement incentives in which eligibility to win will be conditional on medication adherence and registering a weight measurement; and, (4) will determine their preferences for Way to Health platform communication methods during the study.
  Interventions: Behavioral: Support partner; Behavioral: Engagement incentives; Behavioral: Electronic pill bottle; Behavioral: Bluetooth scale

INTERVENTIONS:
Behavioral: Support partner — Participants will identify a support partner who will be contacted if the participant is non-adherent to their diuretic and/or weighing-in.
Behavioral: Engagement incentives — Participants will be entered into a daily lottery, for which their participation is contingent on adhering to their diuretic and to weighing-in on the previous day.
Behavioral: Electronic pill bottle — Participant adherence to their diuretic will be monitored on a daily basis and participants will be contacted if they are non-adherent to this medication.
Behavioral: Bluetooth scale — Participant adherence to stepping on their scale will be monitored on a daily basis and participants will be contacted if they are non-adherent to weighing-in. Participant weight gain will also be monitored, and if weight gain exceeds a specific threshold, the managing physician will be notified through the electronic medical record system. Managing providers will also be sent a weekly report of weight measurements.

SUMMARY:
This study offers remote monitoring devices for weight and medication adherence, combined with behavioral economic approaches, to patients with congestive heart failure (CHF). This pilot study aims to evaluate the feasibility of enrollment processes and intervention roll-out to inform a randomized controlled trial, to estimate the readmission rate of participants, and to assess if and how managing clinicians respond to weight gain alerts entered into a participant's electronic medical record.

DETAILED DESCRIPTION:
The specific aims of this study are: (1) To leverage access to the University of Pennsylvania Health System (UPHS) CHF clinic, PennChart (electronic medical record system) resources for identifying eligible patients, and the Way to Health (WTH) platform to launch a pilot study that will inform a randomized controlled trial; (2) to evaluate the feasibility of the enrollment processes and intervention roll-out to inform a randomized controlled trial; (3) to estimate the readmission rate of participants; and, (4) to assess if and how managing physicians respond to weight gain alerts entered into participant charts in PennChart. In this pilot study, no randomization will occur and all participants will receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Discharged to home within the past 30 days from a UPHS hospital with a principal diagnosis of CHF
* Aged 18 to 80 years old
* Will receive follow-up in a UPHS outpatient clinic by a cardiologist or primary care physician

Exclusion Criteria:

* Less than 18 years old or older than 80 years old
* Will not or cannot provide informed consent
* Have a markedly shortened life expectancy (listed for heart transplant, have ventricular assist device, are inotrope dependent, have metastatic cancer, or have dementia)
* Have end-stage renal disease
* Have a glomerular filtration rate <25 ml/min
* On dialysis
* Heart failure is managed with a CardioMEMS monitor
* Receiving another remote monitoring/telemedicine intervention
* Receiving follow-up care outside of UPHS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of patients successfully setup on the remote monitoring devices | 30 days

SECONDARY OUTCOMES:
All-cause readmission rate | 30 days
Proportion of weight gain alerts that are opened | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; David A Asch, MD, MBA, Principal Investigator — University of Pennsylvania

IPD SHARING:
Plan to Share IPD: No